CLINICAL TRIAL: NCT07390617
Title: Interrogating Enfortumab Vedotin-associated Neuropathy in Patients With Metastatic Urothelial Carcinoma Receiving Enfortumab Vedotin
Brief Title: A Study of Neuropathy Caused by Enfortumab Vedotin in People With Urothelial Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-371
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Neuropathy; Urothelial Carcinoma; Metastatic Urothelial Carcinoma
Keywords: urothelial carcinoma; metastatic urothelial carcinoma; neuropathy; Memorial Sloan Kettering Cancer Center; 25-371
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Urothelial Carcinoma: Participants will have histological or cytologically confirmed urothelial carcinoma
  Interventions: Other: Non-therapeutic Nerve Conduction Studies; Other: Non-therapeutic assessment of patient-reported neuropathy

INTERVENTIONS:
Other: Non-therapeutic Nerve Conduction Studies — Non-invasive nerve conduction studies (NCS) offer an objective, quantitative approach to assess peripheral nerve function, particularly in sensory fibers, which are most commonly affected in chemotherapy-induced peripheral neuropathy/CIPN
Other: Non-therapeutic assessment of patient-reported neuropathy — To evaluate the incidence and severity of chemotherapy-induced peripheral neuropathy (CIPN) in participants receiving enfortumab vedotin, we will collect non-therapeutic, participant-reported outcomes

SUMMARY:
The purpose of this study is to see how results of nerve tests change in people with urothelial cancer who receive treatment with enfortumab vedotin (EV)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by and HIPAA authorization for release of personal health information obtained from the research participant.
* Able to speak and read English to a sufficient level of fluency to provide informed consent and complete the study questionnaires.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 3 within 28 days prior to consent.
* Histological or cytologically confirmed urothelial carcinoma.
* Patients must be planned to start systemic therapy with enfortumab vedotin
* At time of enrollment, patients must be planned to start enfortumab with or without pembrolizumab

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Inability of the subject to understand and comply with study procedures.
* Having previously received enfortumab vedotin
* Students/employees of the study institution, pregnant women, prisoners, and institutionalized individuals (to prevent enrollment of vulnerable subjects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since EV will be given per standard of care, we have not included inclusion criteria relevant to the safety of administering EV itself, since that will be left to the discretion of the treating clinician in a real-world, usual care setting, as is standard practice for non-therapeutic studies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in Nerve Conduction Studies/NCS from baseline to 12-15 weeks | up to 4 months
  Describe change in Nerve Conduction Studies/NCS from baseline to 12-15 weeks. An NCS measures the flow of electrical current through motor and sensory nerves.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lage, MD, MBA, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org